CLINICAL TRIAL: NCT00114972
Title: SYNTAX Study: SYNergy Between PCI With TAXUS and Cardiac Surgery
Brief Title: SYNTAX Study: TAXUS Drug-Eluting Stent Versus Coronary Artery Bypass Surgery for the Treatment of Narrowed Arteries
Acronym: SYNTAX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Cardialysis BV (Industry)
Responsible Party: Nic Van Dyck, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2024; 90169394
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease
Keywords: Three-vessel coronary artery disease; Left main coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass; JCAD protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI with DES (Experimental)
  Interventions: Device: Polymer-based Paclitaxel-Eluting TAXUS Express2-SR Stent
- CABG (coronary artery bypass graft) (Active Comparator): Coronary Artery Bypass Graft
  Interventions: Procedure: Coronary Artery Bypass Surgery

INTERVENTIONS:
Device: Polymer-based Paclitaxel-Eluting TAXUS Express2-SR Stent — Drug Eluting Stent
  Other Names: Percutaneous coronary intervention; Paclitaxel eluting stent; 3 vessel disease; Left main stem
  Arms: PCI with DES
Procedure: Coronary Artery Bypass Surgery — Coronary Artery Bypass Surgery
  Other Names: Coronary artery disease; Coronary artery bypass graft; Left Main coronary artery
  Arms: CABG (coronary artery bypass graft)

SUMMARY:
The SYNTAX trial is designed to determine the best treatment for patients with complex coronary disease (blocked or narrowed arteries in both the right and left sides of the heart) by randomizing patients to receive either percutaneous coronary intervention (PCI) with polymer-based paclitaxel-eluting TAXUS stents or to coronary artery bypass surgery (CABG).

DETAILED DESCRIPTION:
Due to the introduction of drug-eluting stents (DESs) and to improvements in therapy for both percutaneous coronary intervention (PCI) and coronary artery bypass surgery (CABG) patients, PCI is challenging CABG as the gold standard for treatment of three vessel (3VD) and left main (LM) coronary disease.

SYNTAX is a novel, randomized trial with nested registries comparing PCI with paclitaxel-eluting TAXUS stents to CABG for 3VD and LM patients to evaluate the best treatment for these patients with complex coronary disease.

Patients at participating centers will be evaluated by both a cardiothoracic surgeon and by an interventional cardiologist.

Those patients who are determined to be eligible for treatment by both PCI and CABG will be randomized to receive either PCI with a polymer-based paclitaxel-eluting TAXUS stent or CABG.

Patients who are determined to be unsuitable for treatment by PCI will be treated by CABG and will be entered into a CABG registry to help define the patient population in which stenting continues to be an unacceptable treatment option.

Similarly, patients who are determined to be unsuitable for treatment by CABG will be treated by PCI, using any interventional techniques or devices with or without the use of DES, and entered into a PCI registry to help define the patients for whom CABG is considered inappropriate.

ELIGIBILITY:
Inclusion Criteria:

* Three-vessel disease, left main disease or LM equivalent with or without 1, 2 or 3VD (left anterior descending [LAD], left circumflex [LCX], right coronary artery [RCA] territory)
* De novo lesions with at least 50% stenosis
* Myocardial ischemia (stable, unstable, silent)

Exclusion Criteria:

* Prior PCI or CABG
* Acute myocardial infarction (with creatinine kinase >2x upper limit of normal)
* Concomitant cardiac valve disease requiring surgical therapy (reconstruction or replacement)
* Participation or planned participation in another cardiovascular clinical study before 1 year follow-up is completed
* Inability to give informed consent due to mental condition, mental retardation, or language barrier

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Serruys, MD, PhD, Principal Investigator — Erasmus Medical Center; Friedrich W Mohr, MD, Principal Investigator — Heart Center Leipzig - University Hospital; Monika Hanisch, PhD, Study Director — Boston Scientific Corporation
Locations (106):
- United States (32):
  - Mercy General Hospital, Sacramento, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - Munroe Medical Center, Ocala, Florida
  - Ocala Heart Institue, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Evanston Hospital, Evanston, Illinois
  - Rockford Cardiology Research Foundation (St. Anthony's Medical Center), Rockford, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Tufts New England Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Mary's Hospital, Rochester, Minnesota
  - SUNY - Stony Brook School of Medicine, Stony Brook, New York
  - SJH Cardiology Associates, Syracuse, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Cardiovascular and Thoracic Surgeons of Greensboro, Greensboro, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - St. Mary's Medical Center, Langhorne, Pennsylvania
  - Medical City Dallas Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - San Antonio Endovascular Heart Institue, San Antonio, Texas
  - Sentara Norfolk General Hospital 1st Fl, Norfolk, Virginia
- Austria (2):
  - Univ. Klinik für Herzchirurgie Landeskliniken, Salzburg
  - Allgemeines Krankenhaus AKH, Vienna
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Academisch Ziekenhuis Middelheim, Antwerp
  - Universitair Ziekenhuis, Ghent
  - Centre Hôpital Universitaire Sart Tilman, Liège
- Czechia (2):
  - University Hospital Vinohrady, Prague
  - Interni Klinika VFN, Prague
- Skejby Sygehus, Aarhus, Denmark
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - University of Helsinki Meilahti Hospital, Helsinki
- France (7):
  - Clinique St Augustin, Bordeaux
  - Institut Cardiovasculaire Paris Sud - Massy, Massy
  - Clinique Saint-Hilaire Rouen, Rouen
  - Centre Hopital Universitaire Rouen - Hopital Charles Nicolle, Rouen
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Centre Hôpital Universitaire Rangueil, Toulouse
- Germany (12):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Universitatsklinik Charite Berlin, Campus Mitte, Berlin
  - Campus Virchow Klinikum Herzkatheterlabor, Berlin
  - Charite Universitaetsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Campus Kiel, Kiel
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Herzzentrum Universität Leipzig, Leipzig
  - Medizinische Universitaet Luebeck, Lübeck
  - Klinikum Grosshadern, München
  - Krankenhaus der Barmherzigen Brüder, Trier
- Hungary (3):
  - National Medical Center, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Medical School of University PECS, Pécs
- Italy (8):
  - Ospedale Riuniti di Bergamo, Bergamo
  - Istituto di Fisiologia Clinica, Stabilimento di Massa Ospedale, Massa
  - Ospedale San Raffaele, Milan
  - Ospedale Civile di Mirano, Mirano
  - IRCCS Policlinico S. Matteo, Pavia
  - Policlinico San Matteo, Pavia
  - Policlinico Agostino Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano
- P. Stradins University Hospital, Riga, Latvia
- Netherlands (6):
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Academisch Ziekenhuis Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - Erasmus MC - University Medical Center Rotterdam, Rotterdam
  - Isala Klinieken, De Weezenlanden, Zwolle
- Rikshospitalet, Oslo, Norway
- Poland (4):
  - Medical University of Silesia - Katowice, Katowice
  - John Paul II Hospital, Krakow
  - Jagiellonian University of Cardiology, Krakow
  - National Institute of Cardiology, Warsaw
- Hospital de Santa Marta, Lisbon, Portugal
- Spain (5):
  - Hospital General de Alicante, Alicante
  - Hospital General Universitario, Alicante
  - Hospital Clinico Y Provincial, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Salamanca, Salamanca
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital of Lund, Lund
  - Lund University Hospital, Lund
  - Karolinska Universitets Sjukhuset - Stockholm, Stockholm
  - Akademiska sjukhuset, Uppsala
  - University Hospital Uppsala, Uppsala
- United Kingdom (9):
  - Royal Sussex County Hospital, Brighton, East Sussex
  - Western Infirmary, Glasgow
  - Glenfield Hospital, Leicester
  - University Hospitals of Leicester NHS Trust Glenfield Hospital, Leicester
  - London Chest Hospital, London
  - St Thomas Hospital, London
  - King's College Hospital London, London
  - John Radcliffe Infirmary Oxford II, Oxford
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Serruys PW, Ninomiya K, Revaiah PC, Gao C, Garg S, van Klaveren D, Onuma Y, Kappetein AP, Davierwala P, Mack M, Thuijs DJFM, Taggart DP, Milojevic M. Ten-year survival benefit and appropriateness of surgical versus percutaneous revascularization in synergy between percutaneous coronary intervention with Taxus and cardiac surgery randomized trial. Eur J Cardiothorac Surg. 2024 Nov 4;66(5):ezae391. doi: 10.1093/ejcts/ezae391. PMID 39447048
- [Derived] Gaba P, Sabik JF, Murphy SA, Bellavia A, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Christiansen EH, Holm NR, Nielsen PH, Sabatine MS, Stone GW, Bergmark BA. Percutaneous Coronary Intervention Versus Coronary Artery Bypass Grafting in Patients With Left Main Disease With and Without Diabetes: Findings From a Pooled Analysis of 4 Randomized Clinical Trials. Circulation. 2024 Apr 23;149(17):1328-1338. doi: 10.1161/CIRCULATIONAHA.123.065571. Epub 2024 Mar 11. PMID 38465592
- [Derived] Ninomiya K, Kageyama S, Shiomi H, Kotoku N, Masuda S, Revaiah PC, Garg S, O'Leary N, van Klaveren D, Kimura T, Onuma Y, Serruys PW; SYNTAX Investigators. Can Machine Learning Aid the Selection of Percutaneous vs Surgical Revascularization? J Am Coll Cardiol. 2023 Nov 28;82(22):2113-2124. doi: 10.1016/j.jacc.2023.09.818. PMID 37993203
- [Derived] Ninomiya K, Kageyama S, Garg S, Masuda S, Kotoku N, Revaiah PC, O'leary N, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Can machine learning unravel unsuspected, clinically important factors predictive of long-term mortality in complex coronary artery disease? A call for 'big data'. Eur Heart J Digit Health. 2023 Feb 28;4(3):275-278. doi: 10.1093/ehjdh/ztad014. eCollection 2023 May. PMID 37265868
- [Derived] Gaba P, Christiansen EH, Nielsen PH, Murphy SA, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Stone GW, Sabik JF, Sabatine MS, Holm NR, Bergmark BA. Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft Surgery for Left Main Disease in Patients With and Without Acute Coronary Syndromes: A Pooled Analysis of 4 Randomized Clinical Trials. JAMA Cardiol. 2023 Jul 1;8(7):631-639. doi: 10.1001/jamacardio.2023.1177. PMID 37256598
- [Derived] Wang R, Lunardi M, Hara H, Gao C, Ono M, Davierwala PM, Holmes DR, Mohr FW, Curzen N, Burzotta F, van Geuns RJ, Kappetein AP, Head SJ, Thuijs DJFM, Tao L, Garg S, Onuma Y, Wijns W, Serruys PW. Impact of repeat revascularization within 5 years on 10-year mortality after percutaneous or surgical revascularization. Clin Res Cardiol. 2023 Sep;112(9):1302-1311. doi: 10.1007/s00392-023-02211-6. Epub 2023 May 8. PMID 37150783
- [Derived] Ono M, Serruys PW, Kawashima H, Lunardi M, Wang R, Hara H, Gao C, Garg S, O'Leary N, Wykrzykowska JJ, Piek JJ, Holmes DR, Morice MC, Kappetein AP, Noack T, Davierwala PM, Spertus JA, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. Impact of residual angina on long-term clinical outcomes after percutaneous coronary intervention or coronary artery bypass graft for complex coronary artery disease. Eur Heart J Qual Care Clin Outcomes. 2023 Aug 7;9(5):490-501. doi: 10.1093/ehjqcco/qcac052. PMID 36001991
- [Derived] Ono M, Serruys PW, Garg S, Kawashima H, Gao C, Hara H, Lunardi M, Wang R, O'Leary N, Wykrzykowska JJ, Piek JJ, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Noack T, Mohr FW, Davierwala PM, Spertus JA, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. Effect of Patient-Reported Preprocedural Physical and Mental Health on 10-Year Mortality After Percutaneous or Surgical Coronary Revascularization. Circulation. 2022 Oct 25;146(17):1268-1280. doi: 10.1161/CIRCULATIONAHA.121.057021. Epub 2022 Jul 18. PMID 35862109
- [Derived] Ono M, Hara H, Gao C, Kawashima H, Wang R, O'Leary N, Wykrzykowska JJ, Piek JJ, Mack MJ, Holmes D, Morice MC, Head S, Kappetein AP, Noack T, Davierwala PM, Mohr FW, Garg S, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Mortality after multivessel revascularisation involving the proximal left anterior descending artery. Heart. 2022 Oct 28;108(22):1784-1791. doi: 10.1136/heartjnl-2022-320934. PMID 35732441
- [Derived] Ninomiya K, Serruys PW, Garg S, Gao C, Masuda S, Lunardi M, Lassen JF, Banning AP, Colombo A, Burzotta F, Morice MC, Mack MJ, Holmes DR, Davierwala PM, Thuijs DJFM, van Klaveren D, Onuma Y; SYNTAX Extended Survival Investigators. Predicted and Observed Mortality at 10 Years in Patients With Bifurcation Lesions in the SYNTAX Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1231-1242. doi: 10.1016/j.jcin.2022.04.025. Epub 2022 May 17. PMID 35595676
- [Derived] Takahashi K, Serruys PW, Fuster V, Farkouh ME, Spertus JA, Cohen DJ, Park SJ, Park DW, Ahn JM, Onuma Y, Kent DM, Steyerberg EW, van Klaveren D; SYNTAX, BEST, and FREEDOM Trial investigators. External Validation of the FREEDOM Score for Individualized Decision Making Between CABG and PCI. J Am Coll Cardiol. 2022 Apr 19;79(15):1458-1473. doi: 10.1016/j.jacc.2022.01.049. PMID 35422242
- [Derived] Kawashima H, Serruys PW, Hara H, Ono M, Gao C, Wang R, Garg S, Sharif F, de Winter RJ, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year All-Cause Mortality Following Percutaneous or Surgical Revascularization in Patients With Heavy Calcification. JACC Cardiovasc Interv. 2022 Jan 24;15(2):193-204. doi: 10.1016/j.jcin.2021.10.026. Epub 2021 Dec 29. PMID 34973904
- [Derived] Hara H, Kawashima H, Ono M, Takahashi K, Mack MJ, Holmes DR Jr, Morice MC, Davierwala PM, Mohr FW, Thuijs DJFM, Kappetein AP, O'Leary N, van Klaveren D, Onuma Y, Serruys PW. Impact of preprocedural biological markers on 10-year mortality in the SYNTAXES trial. EuroIntervention. 2022 Apr 22;17(18):1477-1487. doi: 10.4244/EIJ-D-21-00415. PMID 34669586
- [Derived] Thuijs DJFM, Davierwala P, Milojevic M, Deo SV, Noack T, Kappetein AP, Serruys PW, Mohr FW, Morice MC, Mack MJ, Stahle LEGE, Verberkmoes NJ, Holmes DR, Head SJ; SYNTAX Extended Survival Investigators. Long-term survival after coronary bypass surgery with multiple versus single arterial grafts. Eur J Cardiothorac Surg. 2022 Mar 24;61(4):925-933. doi: 10.1093/ejcts/ezab392. PMID 34618017
- [Derived] Wang R, Garg S, Gao C, Kawashima H, Ono M, Hara H, van Geuns RJ, Morice MC, Davierwala PM, Kappetein AP, Holmes DR, Wijns W, Tao L, Onuma Y, Serruys PW. Impact of established cardiovascular disease on 10-year death after coronary revascularization for complex coronary artery disease. Clin Res Cardiol. 2021 Oct;110(10):1680-1691. doi: 10.1007/s00392-021-01922-y. Epub 2021 Aug 25. PMID 34432113
- [Derived] Davierwala PM, Gao C, Thuijs DJFM, Wang R, Hara H, Ono M, Noack T, Garg S, O'leary N, Milojevic M, Kappetein AP, Morice MC, Mack MJ, van Geuns RJ, Holmes DR, Gaudino M, Taggart DP, Onuma Y, Mohr FW, Serruys PW; SYNTAX Extended Survival Investigators. Single or multiple arterial bypass graft surgery vs. percutaneous coronary intervention in patients with three-vessel or left main coronary artery disease. Eur Heart J. 2022 Mar 31;43(13):1334-1344. doi: 10.1093/eurheartj/ehab537. PMID 34405875
- [Derived] Wang R, Serruys PW, Gao C, Hara H, Takahashi K, Ono M, Kawashima H, O'leary N, Holmes DR, Witkowski A, Curzen N, Burzotta F, James S, van Geuns RJ, Kappetein AP, Morel MA, Head SJ, Thuijs DJFM, Davierwala PM, O'Brien T, Fuster V, Garg S, Onuma Y. Ten-year all-cause death after percutaneous or surgical revascularization in diabetic patients with complex coronary artery disease. Eur Heart J. 2021 Dec 28;43(1):56-67. doi: 10.1093/eurheartj/ehab441. PMID 34405232
- [Derived] Ono M, Kawashima H, Hara H, Mancone M, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Noack T, Mohr FW, Davierwala PM, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Impact of major infections on 10-year mortality after revascularization in patients with complex coronary artery disease. Int J Cardiol. 2021 Oct 15;341:9-12. doi: 10.1016/j.ijcard.2021.08.013. Epub 2021 Aug 8. PMID 34375706
- [Derived] Kawashima H, Serruys PW, Ono M, Hara H, O'Leary N, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Sharif F, McEvoy JW, Onuma Y; SYNTAX Extended Survival Investigators. Impact of Optimal Medical Therapy on 10-Year Mortality After Coronary Revascularization. J Am Coll Cardiol. 2021 Jul 6;78(1):27-38. doi: 10.1016/j.jacc.2021.04.087. PMID 34210411
- [Derived] Ono M, Serruys PW, Hara H, Kawashima H, Gao C, Wang R, Takahashi K, O'Leary N, Wykrzykowska JJ, Sharif F, Piek JJ, Garg S, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Noack T, Davierwala PM, Mohr FW, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year Follow-Up After Revascularization in Elderly Patients With Complex Coronary Artery Disease. J Am Coll Cardiol. 2021 Jun 8;77(22):2761-2773. doi: 10.1016/j.jacc.2021.04.016. PMID 34082905
- [Derived] Ono M, Kawashima H, Hara H, O'Leary N, Gao C, Wang R, Takahashi K, Wykrzykowska JJ, Piek JJ, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Noack T, Friedrich MW, Davierwala PM, McEvoy JW, Onuma Y, Serruys PW. Impact of Body Composition Indices on Ten-year Mortality After Revascularization of Complex Coronary Artery Disease (From the Syntax Extended Survival Trial). Am J Cardiol. 2021 Jul 15;151:30-38. doi: 10.1016/j.amjcard.2021.04.008. Epub 2021 May 26. PMID 34049676
- [Derived] Takahashi K, Serruys PW, Gao C, Ono M, Wang R, Thuijs DJFM, Mack MJ, Curzen N, Mohr FW, Davierwala P, Milojevic M, Wykrzykowska JJ, de Winter RJ, Sharif F, Onuma Y, Head SJ, Kappetein AP, Morice MC, Holmes DR Jr; SYNTAX Extended Survival Study Investigators. Ten-Year All-Cause Death According to Completeness of Revascularization in Patients With Three-Vessel Disease or Left Main Coronary Artery Disease: Insights From the SYNTAX Extended Survival Study. Circulation. 2021 Jul 13;144(2):96-109. doi: 10.1161/CIRCULATIONAHA.120.046289. Epub 2021 May 20. PMID 34011163
- [Derived] Wang R, Tomaniak M, Takahashi K, Gao C, Kawashima H, Hara H, Ono M, van Klaveren D, van Geuns RJ, Morice MC, Davierwala PM, Mack MJ, Witkowski A, Curzen N, Berti S, Burzotta F, James S, Kappetein AP, Head SJ, Thuijs DJFM, Mohr FW, Holmes DR, Tao L, Onuma Y, Serruys PW. Impact of chronic obstructive pulmonary disease on 10-year mortality after percutaneous coronary intervention and bypass surgery for complex coronary artery disease: insights from the SYNTAX Extended Survival study. Clin Res Cardiol. 2021 Jul;110(7):1083-1095. doi: 10.1007/s00392-021-01833-y. Epub 2021 Mar 12. PMID 33710385
- [Derived] Takahashi K, Thuijs DJFM, Gao C, Ono M, Holmes DR, Mack MJ, Morice MC, Mohr FW, Curzen N, Davierwala PM, Milojevic M, Dawkins KD, Wykrzykowska JJ, de Winter RJ, McEvoy JW, Onuma Y, Head SJ, Kappetein AP, Serruys PW; SYNTAX Extended Survival Study Investigators. Ten-year all-cause mortality according to smoking status in patients with severe coronary artery disease undergoing surgical or percutaneous revascularization. Eur J Prev Cardiol. 2022 Mar 11;29(2):312-320. doi: 10.1093/eurjpc/zwaa089. PMID 33624046
- [Derived] Kawashima H, Takahashi K, Ono M, Hara H, Wang R, Gao C, Sharif F, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Serruys PW, Onuma Y; SYNTAX Extended Survival Investigators. Mortality 10 Years After Percutaneous or Surgical Revascularization in Patients With Total Coronary Artery Occlusions. J Am Coll Cardiol. 2021 Feb 9;77(5):529-540. doi: 10.1016/j.jacc.2020.11.055. PMID 33538250
- [Derived] Wang R, Takahashi K, Garg S, Thuijs DJFM, Kappetein AP, Mack MJ, Morice MC, Mohr FW, Curzen N, Davierwala P, Milojevic M, van Geuns RJ, Head SJ, Onuma Y, Holmes DR Jr, Serruys PW. Ten-year all-cause death following percutaneous or surgical revascularization in patients with prior cerebrovascular disease: insights from the SYNTAX Extended Survival study. Clin Res Cardiol. 2021 Oct;110(10):1543-1553. doi: 10.1007/s00392-020-01802-x. Epub 2021 Jan 30. PMID 33517534
- [Derived] Hara H, Serruys PW, Takahashi K, Kawashima H, Ono M, Gao C, Wang R, Mohr FW, Holmes DR, Davierwala PM, Head SJ, Thuijs DJFM, Milojevic M, Kappetein AP, Garg S, Onuma Y, Mack MJ; SYNTAX Extended Survival Investigators. Impact of Peri-Procedural Myocardial Infarction on Outcomes After Revascularization. J Am Coll Cardiol. 2020 Oct 6;76(14):1622-1639. doi: 10.1016/j.jacc.2020.08.009. PMID 33004127
- [Derived] Hara H, Takahashi K, van Klaveren D, Wang R, Garg S, Ono M, Kawashima H, Gao C, Mack M, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Onuma Y, Noack T, Mohr FW, Davierwala PM, Serruys PW; SYNTAX Extended Survival Investigators. Sex Differences in All-Cause Mortality in the Decade Following Complex Coronary Revascularization. J Am Coll Cardiol. 2020 Aug 25;76(8):889-899. doi: 10.1016/j.jacc.2020.06.066. PMID 32819461
- [Derived] Modolo R, Chichareon P, Kogame N, Dressler O, Crowley A, Ben-Yehuda O, Puskas J, Banning A, Taggart DP, Kappetein AP, Sabik JA, Onuma Y, Stone GW, Serruys PW. Contemporary Outcomes Following Coronary Artery Bypass Graft Surgery for Left Main Disease. J Am Coll Cardiol. 2019 Apr 23;73(15):1877-1886. doi: 10.1016/j.jacc.2018.12.090. PMID 30999989
- [Derived] Milojevic M, Head SJ, Mack MJ, Mohr FW, Morice MC, Dawkins KD, Holmes DR Jr, Serruys PW, Kappetein AP. Influence of practice patterns on outcome among countries enrolled in the SYNTAX trial: 5-year results between percutaneous coronary intervention and coronary artery bypass grafting. Eur J Cardiothorac Surg. 2017 Sep 1;52(3):445-453. doi: 10.1093/ejcts/ezx104. PMID 28520861
- [Derived] Sotomi Y, Onuma Y, Cavalcante R, Ahn JM, Lee CW, van Klaveren D, de Winter RJ, Wykrzykowska JJ, Farooq V, Morice MC, Steyerberg EW, Park SJ, Serruys PW. Geographical Difference of the Interaction of Sex With Treatment Strategy in Patients With Multivessel Disease and Left Main Disease: A Meta-Analysis From SYNTAX (Synergy Between PCI With Taxus and Cardiac Surgery), PRECOMBAT (Bypass Surgery Versus Angioplasty Using Sirolimus-Eluting Stent in Patients With Left Main Coronary Artery Disease), and BEST (Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease) Randomized Controlled Trials. Circ Cardiovasc Interv. 2017 May;10(5):e005027. doi: 10.1161/CIRCINTERVENTIONS.117.005027. PMID 28495897
- [Derived] Abdallah MS, Wang K, Magnuson EA, Osnabrugge RL, Kappetein AP, Morice MC, Mohr FA, Serruys PW, Cohen DJ; SYNTAX Trial Investigators. Quality of Life After Surgery or DES in Patients With 3-Vessel or Left Main Disease. J Am Coll Cardiol. 2017 Apr 25;69(16):2039-2050. doi: 10.1016/j.jacc.2017.02.031. PMID 28427580
- [Derived] Cavalcante R, Sotomi Y, Zeng Y, Lee CW, Ahn JM, Collet C, Tenekecioglu E, Suwannasom P, Onuma Y, Park SJ, Serruys PW. Coronary bypass surgery versus stenting in multivessel disease involving the proximal left anterior descending coronary artery. Heart. 2017 Mar;103(6):428-433. doi: 10.1136/heartjnl-2016-309720. Epub 2016 Sep 20. PMID 27651390
- [Derived] Migliorini A, Valenti R, Parodi G, Vergara R, Buonamici P, Cerisano G, Carrabba N, Antoniucci D. Angiographic and Clinical Outcomes After Everolimus-Eluting Stenting for Unprotected Left Main Disease and High Anatomic Coronary Complexity. JACC Cardiovasc Interv. 2016 May 23;9(10):1001-7. doi: 10.1016/j.jcin.2016.02.016. PMID 27198680
- [Derived] Milojevic M, Head SJ, Parasca CA, Serruys PW, Mohr FW, Morice MC, Mack MJ, Stahle E, Feldman TE, Dawkins KD, Colombo A, Kappetein AP, Holmes DR Jr. Causes of Death Following PCI Versus CABG in Complex CAD: 5-Year Follow-Up of SYNTAX. J Am Coll Cardiol. 2016 Jan 5;67(1):42-55. doi: 10.1016/j.jacc.2015.10.043. PMID 26764065
- [Derived] Osnabrugge RL, Magnuson EA, Serruys PW, Campos CM, Wang K, van Klaveren D, Farooq V, Abdallah MS, Li H, Vilain KA, Steyerberg EW, Morice MC, Dawkins KD, Mohr FW, Kappetein AP, Cohen DJ; SYNTAX trial investigators. Cost-effectiveness of percutaneous coronary intervention versus bypass surgery from a Dutch perspective. Heart. 2015 Dec;101(24):1980-8. doi: 10.1136/heartjnl-2015-307578. Epub 2015 Nov 9. PMID 26552756
- [Derived] Parasca CA, Head SJ, Mohr FW, Mack MJ, Morice MC, Holmes DR Jr, Feldman TE, Colombo A, Dawkins KD, Serruys PW, Kappetein AP; SYNTAX Investigators. The impact of a second arterial graft on 5-year outcomes after coronary artery bypass grafting in the Synergy Between Percutaneous Coronary Intervention With TAXUS and Cardiac Surgery Trial and Registry. J Thorac Cardiovasc Surg. 2015 Sep;150(3):597-606.e2. doi: 10.1016/j.jtcvs.2015.05.010. Epub 2015 May 8. PMID 26055439
- [Derived] Iqbal J, Zhang YJ, Holmes DR, Morice MC, Mack MJ, Kappetein AP, Feldman T, Stahle E, Escaned J, Banning AP, Gunn JP, Colombo A, Steyerberg EW, Mohr FW, Serruys PW. Optimal medical therapy improves clinical outcomes in patients undergoing revascularization with percutaneous coronary intervention or coronary artery bypass grafting: insights from the Synergy Between Percutaneous Coronary Intervention with TAXUS and Cardiac Surgery (SYNTAX) trial at the 5-year follow-up. Circulation. 2015 Apr 7;131(14):1269-77. doi: 10.1161/CIRCULATIONAHA.114.013042. Epub 2015 Feb 24. PMID 25847979
- [Derived] Campos CM, Costa F, Garcia-Garcia HM, Bourantas C, Suwannasom P, Valgimigli M, Morel MA, Windecker S, Serruys PW. Anatomic characteristics and clinical implications of angiographic coronary thrombus: insights from a patient-level pooled analysis of SYNTAX, RESOLUTE, and LEADERS Trials. Circ Cardiovasc Interv. 2015 Apr;8(4):e002279. doi: 10.1161/CIRCINTERVENTIONS.114.002279. PMID 25825008
- [Derived] Zhang YJ, Iqbal J, van Klaveren D, Campos CM, Holmes DR, Kappetein AP, Morice MC, Banning AP, Grech ED, Bourantas CV, Onuma Y, Garcia-Garcia HM, Mack MJ, Colombo A, Mohr FW, Steyerberg EW, Serruys PW. Smoking is associated with adverse clinical outcomes in patients undergoing revascularization with PCI or CABG: the SYNTAX trial at 5-year follow-up. J Am Coll Cardiol. 2015 Mar 24;65(11):1107-15. doi: 10.1016/j.jacc.2015.01.014. PMID 25790882
- [Derived] Cohen DJ, Osnabrugge RL, Magnuson EA, Wang K, Li H, Chinnakondepalli K, Pinto D, Abdallah MS, Vilain KA, Morice MC, Dawkins KD, Kappetein AP, Mohr FW, Serruys PW; SYNTAX Trial Investigators. Cost-effectiveness of percutaneous coronary intervention with drug-eluting stents versus bypass surgery for patients with 3-vessel or left main coronary artery disease: final results from the Synergy Between Percutaneous Coronary Intervention With TAXUS and Cardiac Surgery (SYNTAX) trial. Circulation. 2014 Sep 30;130(14):1146-57. doi: 10.1161/CIRCULATIONAHA.114.009985. Epub 2014 Aug 1. PMID 25085960
- [Derived] Zhang YJ, Iqbal J, Campos CM, Klaveren DV, Bourantas CV, Dawkins KD, Banning AP, Escaned J, de Vries T, Morel MA, Farooq V, Onuma Y, Garcia-Garcia HM, Stone GW, Steyerberg EW, Mohr FW, Serruys PW. Prognostic value of site SYNTAX score and rationale for combining anatomic and clinical factors in decision making: insights from the SYNTAX trial. J Am Coll Cardiol. 2014 Aug 5;64(5):423-32. doi: 10.1016/j.jacc.2014.05.022. PMID 25082573
- [Derived] Head SJ, Davierwala PM, Serruys PW, Redwood SR, Colombo A, Mack MJ, Morice MC, Holmes DR Jr, Feldman TE, Stahle E, Underwood P, Dawkins KD, Kappetein AP, Mohr FW. Coronary artery bypass grafting vs. percutaneous coronary intervention for patients with three-vessel disease: final five-year follow-up of the SYNTAX trial. Eur Heart J. 2014 Oct 21;35(40):2821-30. doi: 10.1093/eurheartj/ehu213. Epub 2014 May 21. PMID 24849105
- [Derived] Morice MC, Serruys PW, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR, Choi JW, Ruzyllo W, Religa G, Huang J, Roy K, Dawkins KD, Mohr F. Five-year outcomes in patients with left main disease treated with either percutaneous coronary intervention or coronary artery bypass grafting in the synergy between percutaneous coronary intervention with taxus and cardiac surgery trial. Circulation. 2014 Jun 10;129(23):2388-94. doi: 10.1161/CIRCULATIONAHA.113.006689. Epub 2014 Apr 3. PMID 24700706
- [Derived] Vranckx P, Kalesan B, Stefanini GG, Farooq V, Onuma Y, Silber S, de Vries T, Juni P, Serruys PW, Windecker S. Clinical outcome of patients with stable ischaemic heart disease as compared to those with acute coronary syndromes after percutaneous coronary intervention. EuroIntervention. 2015 Jun;11(2):171-9. doi: 10.4244/EIJV11I2A31. PMID 24531331
- [Derived] Farooq V, Serruys PW, Bourantas CV, Zhang Y, Muramatsu T, Feldman T, Holmes DR, Mack M, Morice MC, Stahle E, Colombo A, de Vries T, Morel MA, Dawkins KD, Kappetein AP, Mohr FW. Quantification of incomplete revascularization and its association with five-year mortality in the synergy between percutaneous coronary intervention with taxus and cardiac surgery (SYNTAX) trial validation of the residual SYNTAX score. Circulation. 2013 Jul 9;128(2):141-51. doi: 10.1161/CIRCULATIONAHA.113.001803. Epub 2013 Jun 13. PMID 23766350
- [Derived] Mack MJ, Head SJ, Holmes DR Jr, Stahle E, Feldman TE, Colombo A, Morice MC, Unger F, Erglis A, Stoler R, Dawkins KD, Serruys PW, Mohr FW, Kappetein AP. Analysis of stroke occurring in the SYNTAX trial comparing coronary artery bypass surgery and percutaneous coronary intervention in the treatment of complex coronary artery disease. JACC Cardiovasc Interv. 2013 Apr;6(4):344-54. doi: 10.1016/j.jcin.2012.11.010. Epub 2013 Mar 20. PMID 23523456
- [Derived] Farooq V, van Klaveren D, Steyerberg EW, Meliga E, Vergouwe Y, Chieffo A, Kappetein AP, Colombo A, Holmes DR Jr, Mack M, Feldman T, Morice MC, Stahle E, Onuma Y, Morel MA, Garcia-Garcia HM, van Es GA, Dawkins KD, Mohr FW, Serruys PW. Anatomical and clinical characteristics to guide decision making between coronary artery bypass surgery and percutaneous coronary intervention for individual patients: development and validation of SYNTAX score II. Lancet. 2013 Feb 23;381(9867):639-50. doi: 10.1016/S0140-6736(13)60108-7. PMID 23439103
- [Derived] Mohr FW, Morice MC, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR Jr, Morel MA, Van Dyck N, Houle VM, Dawkins KD, Serruys PW. Coronary artery bypass graft surgery versus percutaneous coronary intervention in patients with three-vessel disease and left main coronary disease: 5-year follow-up of the randomised, clinical SYNTAX trial. Lancet. 2013 Feb 23;381(9867):629-38. doi: 10.1016/S0140-6736(13)60141-5. PMID 23439102
- [Derived] Head SJ, Holmes DR Jr, Mack MJ, Serruys PW, Mohr FW, Morice MC, Colombo A, Kappetein AP; SYNTAX Investigators. Risk profile and 3-year outcomes from the SYNTAX percutaneous coronary intervention and coronary artery bypass grafting nested registries. JACC Cardiovasc Interv. 2012 Jun;5(6):618-25. doi: 10.1016/j.jcin.2012.02.013. PMID 22721656
- [Derived] Serruys PW, Farooq V, Vranckx P, Girasis C, Brugaletta S, Garcia-Garcia HM, Holmes DR Jr, Kappetein AP, Mack MJ, Feldman T, Morice MC, Stahle E, James S, Colombo A, Pereda P, Huang J, Morel MA, Van Es GA, Dawkins KD, Mohr FW, Steyerberg EW. A global risk approach to identify patients with left main or 3-vessel disease who could safely and efficaciously be treated with percutaneous coronary intervention: the SYNTAX Trial at 3 years. JACC Cardiovasc Interv. 2012 Jun;5(6):606-17. doi: 10.1016/j.jcin.2012.03.016. PMID 22721655
- [Derived] Arnold SV, Magnuson EA, Wang K, Serruys PW, Kappetein AP, Mohr FW, Cohen DJ; SYNTAX Investigators. Do differences in repeat revascularization explain the antianginal benefits of bypass surgery versus percutaneous coronary intervention?: implications for future treatment comparisons. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):267-75. doi: 10.1161/CIRCOUTCOMES.111.964585. Epub 2012 Apr 10. PMID 22496114
- [Derived] Morice MC, Feldman TE, Mack MJ, Stahle E, Holmes DR, Colombo A, Morel MA, van den Brand M, Serruys PW, Mohr F, Carrie D, Fournial G, James S, Leadley K, Dawkins KD, Kappetein AP. Angiographic outcomes following stenting or coronary artery bypass surgery of the left main coronary artery: fifteen-month outcomes from the synergy between PCI with TAXUS express and cardiac surgery left main angiographic substudy (SYNTAX-LE MANS). EuroIntervention. 2011 Oct 30;7(6):670-9. doi: 10.4244/EIJV7I6A109. PMID 21959312
- [Derived] Cohen DJ, Van Hout B, Serruys PW, Mohr FW, Macaya C, den Heijer P, Vrakking MM, Wang K, Mahoney EM, Audi S, Leadley K, Dawkins KD, Kappetein AP; Synergy between PCI with Taxus and Cardiac Surgery Investigators. Quality of life after PCI with drug-eluting stents or coronary-artery bypass surgery. N Engl J Med. 2011 Mar 17;364(11):1016-26. doi: 10.1056/NEJMoa1001508. PMID 21410370
- [Derived] Mohr FW, Rastan AJ, Serruys PW, Kappetein AP, Holmes DR, Pomar JL, Westaby S, Leadley K, Dawkins KD, Mack MJ. Complex coronary anatomy in coronary artery bypass graft surgery: impact of complex coronary anatomy in modern bypass surgery? Lessons learned from the SYNTAX trial after two years. J Thorac Cardiovasc Surg. 2011 Jan;141(1):130-40. doi: 10.1016/j.jtcvs.2010.07.094. PMID 21168023
- [Derived] Morice MC, Serruys PW, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR, Torracca L, van Es GA, Leadley K, Dawkins KD, Mohr F. Outcomes in patients with de novo left main disease treated with either percutaneous coronary intervention using paclitaxel-eluting stents or coronary artery bypass graft treatment in the Synergy Between Percutaneous Coronary Intervention with TAXUS and Cardiac Surgery (SYNTAX) trial. Circulation. 2010 Jun 22;121(24):2645-53. doi: 10.1161/CIRCULATIONAHA.109.899211. Epub 2010 Jun 7. PMID 20530001
- [Derived] Banning AP, Westaby S, Morice MC, Kappetein AP, Mohr FW, Berti S, Glauber M, Kellett MA, Kramer RS, Leadley K, Dawkins KD, Serruys PW. Diabetic and nondiabetic patients with left main and/or 3-vessel coronary artery disease: comparison of outcomes with cardiac surgery and paclitaxel-eluting stents. J Am Coll Cardiol. 2010 Mar 16;55(11):1067-75. doi: 10.1016/j.jacc.2009.09.057. Epub 2010 Jan 14. PMID 20079596
- [Derived] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612

RESULTS

PARTICIPANT FLOW:
Groups:
- CABG: Coronary Artery By-pass Graft (CABG)
- PCI With DES: Percutaneous coronary intervention (PCI) using TAXUS Express Drug Eluting Stent (DES)
Period: Overall Study
Arm/Group | CABG | PCI With DES
Started | 897 | 903
Completed | 849 | 891
Not Completed | 48 | 12
Not completed — Withdrawal by Subject | 40 | 7
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CABG | PCI With DES | Total
Number analyzed (Participants) | 897 | 903 | 1800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 400 | 397 | 797.0
  >=65 years | 497 | 506 | 1003.0
Age Continuous [Mean (Standard Deviation); unit: years] | 64.96 (9.79) | 65.23 (9.66) | 65.09 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 213 | 402
  Male | 708 | 690 | 1398
Region of Enrollment [Number; unit: participants]
  United States | 122 | 123 | 245.0
  Portugal | 7 | 6 | 13.0
  Finland | 12 | 12 | 24.0
  Spain | 26 | 27 | 53.0
  Austria | 24 | 28 | 52.0
  United Kingdom | 132 | 135 | 267.0
  Italy | 96 | 101 | 197.0
  France | 105 | 103 | 208.0
  Hungary | 39 | 44 | 83.0
  Czech Republic | 20 | 20 | 40.0
  Poland | 33 | 33 | 66.0
  Belgium | 47 | 44 | 91.0
  Denmark | 15 | 17 | 32.0
  Norway | 4 | 4 | 8.0
  Latvia | 20 | 20 | 40.0
  Netherlands | 74 | 74 | 148.0
  Germany | 93 | 86 | 179.0
  Sweden | 28 | 26 | 54.0
Angina [Number; unit: participants] — number of particpiants with stable, unstable, or no angina at baseline
  participants
    Participants with Stable Angina at Baseline | 513 | 514 | 1027.0
    Participants with Unstable Angina at Baseline | 251 | 261 | 512.0
    Participants with Silent Ischemia at Baseline | 74 | 74 | 148.0
    Participants with No Angina at Baseline | 59 | 54 | 113.0
Bifurcation lesion (per participant) [Number; unit: participants] — Number of participants with at least one bifurcation lesion as determined by the angiographic core laboratory on the baseline angiogram
  participants
    One or more Bifurcated Lesion(s) | 652 | 649 | 1301.0
    No Bifurcated Lesions | 245 | 254 | 499.0
Blood pressure ≥130/85 mmHg [Number; unit: participants] — number of participants with blood pressure equal or higher than 130/85mmHg
  participants
    Blood Pressure >= 130/85 mmHG | 574 | 622 | 1196.0
    Blood Pressure <130/85 mmHG | 323 | 281 | 604.0
Carotid artery disease [Number; unit: participants] — number of particpants with diagnosed carotid artery disease at baseline
  participants
    Diagnosed Carotid Artery Disease at Baseline | 75 | 73 | 148.0
    No Diagnosed Carotid Artery Disease at Baseline | 822 | 830 | 1652.0
Congestive heart failure [Number; unit: participants] — number of particpants with congestive heart failure at baseline
  participants
    Congestive Heart Failure at Baseline | 47 | 36 | 83.0
    No Congestive Heart Failure at Baseline | 850 | 867 | 1717.0
Current smoking [Number; unit: participants] — Number of participants that were smoking at baseline
  participants
    Smokers at Baseline | 196 | 167 | 363.0
    Non-Smokers at Baseline | 701 | 736 | 1437.0
Diabetes [Number; unit: participants] — All participants with diagnosed diabetes at baseline
  participants
    Diagnosed Diabetes at Baseline | 256 | 255 | 511.0
    No Diagnosed Diabetes at Baseline | 641 | 648 | 1289.0
HDL cholesterol (<40 Male or <50 Female) [Number; unit: participants] — number of male participants with a high-density lipoprotein (HDL)<40 and female particpants with a HDL<50 determined by the central chemistry laboratory
  participants
    Participant HDL Less Than Limit at Baseline | 404 | 379 | 783.0
    Participant HDL Greater Than Limit at Baseline | 493 | 524 | 1017.0
Hyperlipidemia [Number; unit: participants] — participants with hyperlipidemia at baseline
  participants
    Participants with Hyperlipidemia at Baseline | 686 | 705 | 1391.0
    Participants without Hyperlipidemia at Baseline | 211 | 198 | 409.0
Insulin requiring diabetes [Number; unit: participants] — Number of participants with diabetes treated with insulin
  participants
    Participants with Insulin dependent Diabetes | 93 | 89 | 182.0
    Participants with non-Insulin independent Diabetes | 163 | 166 | 329.0
    Nondiabetic Participants | 641 | 648 | 1289.0
Medically treated Diabetes [Number; unit: Participants] — Number of participants with medically treated diabetes.Excludes participants with diabetes treated with diet only.
  Participants
    Diabetic Participants Medically Treated | 221 | 231 | 452.0
    Diabetic Participants Treated through Diet only | 35 | 24 | 59.0
    Non-Diabetic Participants | 641 | 648 | 1289.0
Metabolic Syndrome [Number; unit: participants] — number of participants that met the criteria of metabolic syndrome defined by the American Heart Association
  participants
    Participants with a Metabolic Syndrome | 317 | 339 | 656.0
    Participants without a Metabolic Syndrome | 580 | 564 | 1144.0
Poor LVEF [Number; unit: participants] — number of participants with left ventricular ejection fraction <30% at baseline
  participants
    LVEF <30% at Baseline | 22 | 12 | 34.0
    LVEF >=30% at Baseline | 875 | 891 | 1766.0
Prior MI [Number; unit: participants] — Number of participants who had a myocardial infarction before baseline
  participants
    Myocardial Infarction Before Baseline | 300 | 285 | 585.0
    No Myocardial Infarction Before Baseline | 597 | 618 | 1215.0
Prior Stroke [Number; unit: participants] — number of participants who had a stroke before baseline
  participants
    Stroke Prior to Baseline | 43 | 35 | 78.0
    No Stroke Prior to Baseline | 854 | 868 | 1722.0
Prior TIA [Number; unit: participants] — number of partipants who had a Transient Ischemic Attack before baseline
  participants
    Transient Ischemic Attack Before Baseline | 45 | 39 | 84.0
    No Transient Ischemic Attack before baseline | 852 | 864 | 1716.0
Total Occlusion (per patient) [Number; unit: participants] — Number of participants with at least one total occlusion as determined by the angiografic core laboratory on the baseline angiogram
  participants
    Participants with at least One Total Occlusion | 198 | 217 | 415.0
    Participants with Partial Occlusion(s) | 699 | 686 | 1385.0
Triglyceride levels ≥150 mg/dL [Number; unit: participants] — participants with Triglyceride levels ≥150 mg/dL as determined by a central chemistry laboratorium at baseline
  participants
    Participants with Triglyceride Levels >= 150 mg/dL | 304 | 275 | 579.0
    Participants with Triglyceride Levels <150 mg/dL | 593 | 628 | 1221.0
Additive Euroscore [Mean (Standard Deviation); unit: units on a scale] — Additive EuroSCORE is a prognostic scoring system calculating predicted operative mortality for patients undergoing cardiac surgery; it has been the most rigorously evaluated scoring system in cardiac surgery. A predetermined weighted score is assigned for specified patient-, cardiac-, and operation-related factors; for example, pulmonary hypertension is assigned a score of 2. The sum of scores is the additive EuroSCORE. EuroSCORE is calculated from site reported baseline data. A score of greater than 6 is considered as being predictive of an increased mortality risk. (www.euroscore.org)
  units on a scale | 3.79 (2.69) | 3.75 (2.62) | 3.77 (2.66)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index calculated from participants heigth and weight.
  kg/m2 | 27.91 (4.54) | 28.11 (4.80) | 28.01 (4.67)
Number of lesions per partipant [Mean (Standard Deviation); unit: Number of lesions/Participant] — Average number of lesions per participant as determined by the investigator
  Number of lesions/Participant | 3.99 (1.7) | 3.94 (1.66) | 3.97 (1.68)
Parsonnet Score [Mean (Standard Deviation); unit: units on a scale] — The first scoring system in cardiac surgery to calculate mortality risk and to become popular was the Parsonnet risk stratification system, which was developed in the United States in the 1980s. A predetermined weighted score is assigned for several specified patient-, cardiac-, and operation-related factors; for example, dialysis is assigned a score of 10. A score of greater than 15 is considered as being predictive of an increased mortality risk. Parsonette score is calculated from baseline information.
  units on a scale | 8.43 (6.84) | 8.53 (6.95) | 8.48 (6.9)
Total Syntax Score [Mean (Standard Deviation); unit: units on a scale] — The SYNTAX score characterizes the coronary vasculature. It combines the importance of a diseased coronary artery segment (Leaman score), adverse characteristics of a lesion (ACC/AHA lesion classification) and the modified Duke/ICPS classification for bifurcation lesions. Higher SYNTAX scores are indicative of more complex lesions and disease; thus higher scores would predict worse short-term outcomes. Calculated from angiographic corelab analysis of baseline angiogram. (www.syntaxscore.com)
  units on a scale | 29.1 (11.37) | 28.39 (11.46) | 28.7 (11.42)

OUTCOME MEASURES:

1. Primary Outcome: Primary Clinical Endpoint of 12-Month Binary MACCE.
Description: Number of participants at primary clinical endpoint of 12-Month binary MACCE. MACCE is defined as: all cause death, cerebrovascular event (stroke), cocumented myocardial infarction, repeat revascularization (PCI and/or CABG).
Time Frame: 12 months post enrollment
Population: ITT analysis. Number of participants analyzed equals number of subjects who completed Overall Study, as listed in Participant Flow.
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
participants | 105 | 159

2. Primary Outcome: 12-month Composite Safety Endpoint.
Description: Number of participants at 12-month composite safety endpoint. Composite safety endpoint combines: all cause death, cerebrovascular event (stroke), and documented myocardial infarction.
Time Frame: 12 months after enrollment
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
participants | 65 | 68

3. Secondary Outcome: Overall MACCE at 1 Month Post-procedure and at 6 Months, 3 Years, and 5 Years Post-allocation.
Description: Number of participants with Overall MACCE at 1 month post-procedure and at 6 months, 3 years, and 5 years post-allocation.
Time Frame: 1 month after procedure and 6 months, 3 years, and 5 years post allocation
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
participants
  MACCE 1 month post procedure | 45 | 54
  MACCE 6 months post procedure | 85 | 111

4. Secondary Outcome: Individual Components of MACCE at 1 Month Post-procedure.
Description: Number of participants with individual components of MACCE at 1 month post-procedure. The individual components of MACCE are: all cause death, stroke, documented myocardial infarction, repeat revascularization.
Time Frame: 1 month after procedure
Population: ITT analysis
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 866 | 895
participants
  All cause death | 10 | 20
  Stroke | 9 | 2
  Documented MI | 21 | 31
  Any repeat revascularization | 15 | 31

5. Secondary Outcome: Individual Components of MACCE at 6 Months Post-allocation.
Description: Number of participants with individual components of MACCE at 6 months post-allocation. The individual components of MACCE are: all cause death, stroke, documented myocardial infarction, repeat revascularization.
Time Frame: 6 months post allocation
Population: ITT analysis
Measure: Number; unit: Participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 860 | 893
Participants
  All cause death | 24 | 31
  Stroke | 13 | 2
  Documented MI | 27 | 40
  Any repeat revascularization | 35 | 78

6. Secondary Outcome: Individual Components of MACCE at 1 Year Post-allocation.
Description: Number of participants with individual components of MACCE at 1 year post-allocation. The individual components of MACCE are: all cause death, stroke, documented myocardial infarction, repeat revascularization.
Time Frame: 1 year post allocation
Population: ITT analysis
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
participants
  Death any cause | 30 | 39
  Stroke | 19 | 5
  Documented MI | 28 | 43
  Any repeat revascularization | 50 | 120

7. Secondary Outcome: Freedom From MACCE and Its Components at 1 Year Post-allocation.
Description: Number of participants with freedom from MACCE and its components at 1 year post-allocation. Freedom from MACCE is defined as no MACCE nor any of the individual components of MACCE (all cause death, stroke, documented myocardial infarction, repeat revascularization).
Time Frame: 1 year post allocation
Measure: Number; unit: participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
participants
  Freedom from any MACCE | 744 | 732
  Freedom from any cause death | 819 | 852
  Freedom from stroke | 830 | 886
  Freedom from documented MI | 821 | 848
  Freedom from any repeat revascularization | 799 | 771

8. Secondary Outcome: Freedom From MACCE and Its Components at 3 Years Post-allocation
Time Frame: 3 years post allocation
Reporting Status: Not Posted
Measure: Number; unit: participants

9. Primary Outcome: Repeat Revascularization (PCI and/or CABG).
Description: Number of participants with repeat revascularization (PCI and/or CABG).
Time Frame: 12 Months post enrollment
Measure: Number; unit: Participants
Arm/Group | CABG | PCI With DES
Number analyzed (Participants) | 849 | 891
Participants | 50 | 120

10. Secondary Outcome: Freedom From MACCE and Its Components at 5 Years Post-allocation
Time Frame: 5 years post allocation
Reporting Status: Not Posted
Measure: Number; unit: participants

11. Secondary Outcome: Quality of Life at 1 Month Post-procedure and at 6 Months, 1, 3 and 5 Years Post-allocation
Time Frame: 1 month after procedure and 6 months, 1, 3 and 5 years post allocation
Reporting Status: Not Posted

12. Secondary Outcome: Cost and Cost-effectiveness at 1, 3 and 5 Years Post-allocation
Time Frame: 1 year, 3 and 5 years post allocation
Reporting Status: Not Posted

13. Secondary Outcome: The Characteristics (Including Co-morbidity and Coronary Vascular Lesion Complexity Scoring Referred to as the SYNTAX Score) of the Following: PCI Versus CABG Randomized Cohort, PCI Registry Cohort (CABG Ineligible), CABG Registry Cohort (PCI Ineligible)
Time Frame: 5 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CABG | PCI With DES
Serious Adverse Events (participants affected / at risk) | 391/897 | 357/903
Other Adverse Events (participants affected / at risk) | 509/897 | 405/903
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CABG (N=897) | PCI With DES (N=903)
Abnormal blood test values (Investigations) | 14 (15) | 18 (19) — Total of all abnormal blood tests (increased or decreased) and abnormal diagnostic procedures. Occurrence of each individual event term is less than 1%.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 27 (31) | 20 (20)
Anaphylactic shock , reaction and drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) — Total of events related to immune system disorder like anaphylactic reaction or shock and drug hypersensitivity. Occurrence of each individual event term is less than 1%.
Angina Pectoris (Cardiac disorders) | 30 (49) | 74 (95)
Angina Unstable (Cardiac disorders) | 30 (38) | 66 (85)
Arrhythmia, other rare cardiac disorders (Cardiac disorders) | 51 (58) | 82 (99) — Rare cardiac disorders like ventricular arrhytmias, atrioventricular blocks, cardiomyopathy, valve disease, coronary artery dissection and occlusion. Occurrence of each individual event term is less than 1%.
Atrial Fibrillation (Cardiac disorders) | 45 (47) | 10 (14)
Atrial Flutter (Cardiac disorders) | 10 (11) | 2 (2)
Basedow's Disease (Endocrine disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (8) | 13 (13)
Cardiac Arrest (Cardiac disorders) | 11 (11) | 15 (15)
Cardiac Failure (Cardiac disorders) | 12 (14) | 7 (7)
Cardiac Failure Congestive (Cardiac disorders) | 12 (14) | 7 (8)
Cardiac enzymes increased (Investigations) | 3 (3) | 10 (10)
Cardiac tamponade (Cardiac disorders) | 10 (14) | 3 (4)
Cardiogenic Shock (Cardiac disorders) | 3 (3) | 14 (15)
Carotid artery stenosis (Nervous system disorders) | 9 (9) | 2 (3)
Cataract, lens disorder, renal detachment (Eye disorders) | 3 (4) | 3 (4)
Catheter site haematoma (General disorders) | 1 (1) | 11 (11)
Coronary Artery Thrombosis (Cardiac disorders) | 2 (2) | 28 (41)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 12 (13) | 12 (12)
Hepatobiliary disorders (Hepatobiliary disorders) | 7 (7) | 3 (3) — Total of hepatobiliary disorders like bile duct stone, cholecystitis, hepatic failure and hepatic function abnormal.Occurrence of each individual event term is less than 1%.
Infection and abcess (Infections and infestations) | 44 (45) | 27 (27) — Total of any other infection or abcess. Occurrence of each individual event term is less than 1%.
Injury and procedural complications (Injury, poisoning and procedural complications) | 33 (35) | 15 (16) — Total of all other procedural complications and injuries. Occurrence of each individual event term is less than 1%.
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 12 (12) | 6 (6) — Total of all metabolism and nutrition disorders like hyper- and hypoglycaemie, hypokalaemia, hyponatraemia, dehydration, etc. Occurrence of each individual event term is less than 1%.
Musculoskeletal and connective tissue diorders (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12) — Total of musculoskeletal and connective tissue disorders. Occurrence of each individual event term is less than 1%.
Myocardial Ischaemia (Cardiac disorders) | 2 (2) | 18 (19)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 14 (14) — Total of neoplasms, benign, malignant and unspecified. Occurrence of each individual event term is less than 1%.
Nervous system disorder (Nervous system disorders) | 23 (25) | 13 (13) — Total of all other nervous system disorders. Occurrence of each individual event term is less than 1%.
Non-cardiac chest pain (General disorders) | 6 (6) | 14 (19)
Other gastrointestinal disorders (Gastrointestinal disorders) | 21 (24) | 11 (12) — Sum of all other gastrointestinal disorders like ulcers, pain, hernia, obstructions, vomiting, nausea, etc. Occurrence of each individual event term is less than 1%.
Other general disorders and administration site conditions (General disorders) | 27 (28) | 26 (26) — Other general disorders mainly related to catheter site events like pain, haemorrhage and pyrexia, multi-organ failure, wound healing problems. Occurrence of each individual event term is less than 1%.
Pericardial Effusion (Cardiac disorders) | 10 (11) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 (33) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 9 (9) | 1 (1)
Prostatic disorders (Reproductive system and breast disorders) | 6 (7) | 1 (1) — Total of all reproductive system and breast disorders. All events in this system were related to prostatic disorders. Occurrence of each individual event term is less than 1%.
Psychiatric disorders (Psychiatric disorders) | 12 (12) | 3 (3) — Total of all psychiatric disorders. Occurrence of each individual event term is less than 1%.
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Renal and urinary disorders (Renal and urinary disorders) | 13 (15) | 13 (13) — Total of all other renal and urinary disorders. Occurrence of each individual event term is less than 1%.
Renal failure acute (Renal and urinary disorders) | 22 (23) | 9 (9)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 20 (20) — Total of all other respiratory, thoracic and mediastinal disorders. Occurrence of each individual event term is less than 1%.
Sepsis (Infections and infestations) | 9 (11) | 6 (7)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 0 (0) — Total of surgical and medical procedures. Occurrence of each individual event term is less than 1%.
Vascular disorders (Vascular disorders) | 45 (48) | 48 (48) — Total of vascular disorders. Occurrence of each individual event term is less than 1%.
Vascular graft occlusion (Injury, poisoning and procedural complications) | 28 (29) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 30 (33) | 1 (1)
coagulopathy, iron deficiency anaemia, leukocytosis, thrombocyopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) — Total of other events and subjects affected with these events in this organ system. Event terms are coagulopathy, iron deficiency anaemia, leukocytosis and thrombocyopenia. Occurrence of each individual event term is less than 1%.
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) — Total of skin and subcutaneous tissue disorders. Occurrence of each individual event term is less than 1%.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CABG (N=897) | PCI With DES (N=903)
Anaemia (Blood and lymphatic system disorders) | 104 (109) | 23 (24)
Angina pectoris (Cardiac disorders) | 26 (28) | 61 (70)
Atrial fibrillation (Cardiac disorders) | 123 (129) | 25 (28)
Incision site complication (Injury, poisoning and procedural complications) | 47 (52) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 54 (55) | 2 (2)
Wound infection (Infections and infestations) | 56 (58) | 2 (2)
All other Adverse Events (General disorders) | 509 (1099) | 405 (854) — Total of all other adverse events with an occurrence below the 5% treshold.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days